CLINICAL TRIAL: NCT04098965
Title: Treatment of Scarring and Dysfunction of the Pelvic Floor in Postpartum, Through Physical Therapy or by Medical Recommendations in Consultation
Brief Title: Treatment of Scars and Dysfunctions of the Pelvic Floor in Postpartum
Acronym: NoRFor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, MARÍA DEL PILAR VIDALES COLINAS, Principal Investigator, Universidad de León
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 321311: FISIOTERAPIA
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Physical Therapy Techniques
  Interventions: Other: Pysiotherapy techniques
- Control (Other): physician treatment
  Interventions: Other: physician treatment

INTERVENTIONS:
Other: Pysiotherapy techniques — manual therapy techniques, postural re-education and muscle strengthening
  Arms: Experimental
Other: physician treatment — hygienic-dietary recommendations, Kegel exercises and pain relievers
  Arms: Control

SUMMARY:
Recruitment of patients who have suffered third- and fourth-degree perineal tear during childbirth, and who have given birth at the Hospital Universitario Marqués de Valdecilla (Santander, Spain). They are distributed randomly in two groups an experimental group who apply techniques of physiotherapy and a control group, receiving medical treatment.

At the same time is recruited the same number of patients who have not suffered tear and whose birth has been instrumental, dividing into two groups, control and experimental. And the same number of patients who have given birth but have not suffered tear or instrumental delivery, divided also into control group and experimental.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have dysfunctions in the pelvic floor after childbirth
* Patients who have given birth at the Hospital Universitario Marqués de Valdecilla
* Patients who do not have any medical alteration that does not indicate the treatment

Exclusion Criteria:

* Patients who do not have pelvic floor dysfunctions after childbirth
* Patients who have not given birth at the Hospital Universitario Marqués de Valdecilla
* Patients who have any medical changes that counter the treatment

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
change in VAS from the start to the end | in the begining, at thirth month, at sixth month and at the finish (one year later)
  Pain
Change in SF36 from de start to the end | in the begining, at thirth month, at sixth month and at the finish (one year later)
  quality of life sorth form
Change in EPIQ from de start to the end | in the begining, at thirth month, at sixth month and at the finish (one year later)
  Epidemiology of Prolapse and Incontinence Questionnaire
Change in OXFORD from the start to the end | in the begining, at thirth month, at sixth month and at the finish (one year later)
  muscle strength

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sierrallana, Torrelavega, Cantabria, Spain